CLINICAL TRIAL: NCT05425368
Title: Clinical and Radiographic Evaluation of Silver Diamine Fluoride Versus Mineral Trioxide Aggregate as Indirect Pulp Capping Agents in Deeply Carious Young Permanent Molars Randomized Controlled Clinical Trial
Brief Title: Comparing Two Indirect Pulp Capping Agents for Permanent Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Ahmed Zaghloul, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Indirect pulp capping
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Deep Caries
Keywords: partial caries removal; indirect pulp capping; fluorides
MeSH Terms: interventions — silver diamine fluoride; mineral trioxide aggregate; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Two blinded (patient, radiographic assessor of results)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- silver diamine fluoride group (Experimental): partial caries removal will be carried out then Silver Diamine Fluoride will be applied as indirect pulp capping agent and rubbed for 1 minute followed by Glass ionomer filling
  Interventions: Drug: Silver diamine fluoride
- mineral trioxide aggregate group (Active Comparator): partial caries removal will be carried out then mineral trioxide aggregate will be placed as indirect pulp capping agent followed by glass ionomer filling
  Interventions: Drug: Mineral trioxide aggregate

INTERVENTIONS:
Drug: Silver diamine fluoride — First permanent molars in this group will receive 38% silver diamine fluoride as an indirect pulp capping material.
  Other Names: SDF
  Arms: silver diamine fluoride group
Drug: Mineral trioxide aggregate — First permanent molars in this group will receive mineral trioxide aggregate as an indirect pulp capping material.
  Other Names: MTA
  Arms: mineral trioxide aggregate group

SUMMARY:
Aim of the study:

To evaluate clinical and radiographic success rates of silver diamine fluoride versus mineral trioxide aggregate as indirect pulp capping agents in deeply carious young first permanent molars.

DETAILED DESCRIPTION:
Indirect pulp treatment has become a common maneuver in vital pulp therapy in recent years and is a procedure performed in teeth with deep carious lesions approximating the pulp but without any signs or symptoms of irreversible pulpal changes.

Silver Diamine Fluoride is used to arrest caries lesions in primary teeth but according to the AAPD,2021 more research is needed on the use of SDF to arrest caries lesions in permanent teeth.

ELIGIBILITY:
Inclusion Criteria:

* Patient and parent showing cooperation and compliance.
* Children 9-14 years old
* Vital deeply carious young first permanent molar(s) with complete root formation
* Asymptomatic teeth or without clinical symptoms of spontaneous pain
* Both genders will be included.

Exclusion Criteria:

* Children unable to return for recall visits.
* Any clinical signs of irreversible pulpitis or pulp necrosis (spontaneous pain, pain on percussion, abscess, sinus).
* Any radiographic sign of irreversible pulp pathologies or pulp necrosis (periapical radiolucency, internal or external root resorption)

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dentin bridge formation | 6 months
  Dentin bridge formation will be measured in millimeters on standardized digital radiographs taken by Digital Radiographic examination

SECONDARY OUTCOMES:
Postoperative pain | 1 week
  Postoperative pain will be assessed by questioning the patient or the guardian whether there is postoperative pain or not, Binary (yes or no)
Absence of sinus or fistula | 3 months
  Intraoral Visual examination will be carried out to assess if there is a sinus or fistula, Binary (present/absent)
Absence of sinus or fistula | 6 months
  Intraoral Visual examination will be carried out to assess if there is a sinus or fistula, Binary (present/absent)
radiographic success | 6 months
  Absence of any adverse radiographic findings (Periodontal membrane space widening, bone resorption, pulp stones will be assessed if present or absent by digital radiographic examination, Binary (present or absent)

CONTACTS AND LOCATIONS:
Overall Officials: Manal Ahmed El Sayed, Principal Investigator — Professor of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University; Randa Youssef Abd Al Gawad, Principal Investigator — Professor of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University